CLINICAL TRIAL: NCT00004761
Title: Establishment of the National Epidermolysis Bullosa Registry
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Rockefeller University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Other Study IDs: 199/11706; RU-0170195
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-07

CONDITIONS: Epidermolysis Bullosa
Keywords: dermatologic disorders; epidermolysis bullosa; genetic diseases and dysmorphic syndromes; rare disease
MeSH Terms: conditions — Epidermolysis Bullosa; Skin Diseases; Genetic Diseases, Inborn; Rare Diseases

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Other

SUMMARY:
OBJECTIVES: I. Develop a large roster of well-characterized patients with various forms of inherited and acquired epidermolysis bullosa (EB).

II. Generate a large data bank of clinical, historical, and genetic information concerning these patients.

III. Accumulate donated tissue specimens, including selected cells and DNA, from selected patient subsets for the establishment of permanent tissue cell banks.

IV. Promote and facilitate research in EB.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients are enrolled by mail or clinic visit at 1 of 4 clinical centers. Clinical, epidemiological, and laboratory data are collected.

Medical and family histories are obtained in a detailed interview in person, by phone, or by mail. Diagnostic studies to confirm the type of epidermolysis bullosa are performed as indicated. A pedigree chart is completed on the first affected family member entered.

Selected patients are followed at least biannually. A study duration of approximately 10 years is anticipated.

ELIGIBILITY:
* Clinical diagnosis of epidermolysis bullosa

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1986-09

CONTACTS AND LOCATIONS:
Overall Officials: James G. Krueger, Study Chair — Rockefeller University

REFERENCES:
- [Background] Lin AN, Carter DM: Epidermolysis Bullosa: Basic and Clinical Aspects. New York: Springer Verlag, 1992.